CLINICAL TRIAL: NCT05479227
Title: Bile Duct Injuries During Laparoscopic Cholecystectomies: An 11-year Population-based Study
Status: Completed | Type: Observational
Sponsor: North Estonia Medical Centre (Other)
Collaborators: University of Tartu (Other)
Responsible Party: Principal Investigator, Arvo Reinsoo, Principal investigator, general surgeon, MD, North Estonia Medical Centre
Other Study IDs: AR
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Bile Duct Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with bile duct injuries during laparoscopic cholecystectomy: The data concerning 241 patients´ BDI emergence, severity, management, and outcomes was analyzed
  Interventions: Procedure: Management of bile duct injury

INTERVENTIONS:
Procedure: Management of bile duct injury — There are different options for BDI management, we analyzed their utilization and results

SUMMARY:
The aim of this retrospective study is to review the annual incidence, management, and outcomes of bile duct injuries (BDI) during laparoscopic cholecystectomy (LC) in a population-based cohort during 2008-2018 in Estonia.

DETAILED DESCRIPTION:
The aim of this retrospective study is to review the annual incidence, management, and outcomes of bile duct injuries (BDI) during laparoscopic cholecystectomy (LC) in a population-based cohort during 2008-2018 in Estonia.

Background Data: Iatrogenic bile duct injuries (BDI) following laparoscopic cholecystectomy (LC) result in major morbidity and incidental mortality. There is a lack of unselected population-based cross-sectional studies on the incidence, management, and outcomes of BDI. We hypothesised that due to improved imaging capabilities and collective laparoscopic experience, the BDI incidence will decrease over the study period and compare favourably with contemporary literature.

After IRB approval, all cholecystectomies performed at national public healthcare facilities between 2008 and 2018 were retrospectively reviewed. BDIs were classified according to the Strasberg classification. We hypothesized that due to improved imaging capabilities and collective laparoscopic experience the BDI incidence will decrease over the study period and compare favourably to contemporary literature.

ELIGIBILITY:
Inclusion Criteria:

* all patients with BDI during laparoscopic cholecystectomy (LC)

Exclusion Criteria:

* The sole exclusion criterion in the case selection was cholecystectomy performed primarily using the open method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of patients who experienced a bile duct injury during laparoscopic cholecystectomy during 2008-2018 in Estonian national health care facilities. The data was obtained according to coding in National Health Insurance Fund electronic database. Data on readmissions related to BDIs and their subsequent complications were collected from the National Institute for Health Development repository.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
incidence of bile duct injuries | During the years 2008-2018
  We aimed to review the annual incidence of bile duct injuries in a population-based cohort in Estonia.

CONTACTS AND LOCATIONS:
Overall Officials: Arvo Reinsoo, MD, Principal Investigator — North Estonia Medical Centre
Locations (1):
- Arvo Reinsoo, Tallinn, Estonia

IPD SHARING:
Plan to Share IPD: Undecided